CLINICAL TRIAL: NCT05828329
Title: Virtual Reality to Cope With Academic Exams: Effects on Stress and Academic Performance in Physiotherapy and Nursing Students of University of the Balearic Islands
Brief Title: Virtual Reality to Cope With Academic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IB4958/22PI
Record Dates: First submitted 2023-03-29; First posted 2023-04-25 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stress, Physiological; Stress, Psychological
Keywords: Education; Virtual Reality; Students
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned with a code with which investigators and outcomes assessors will not be able to know from whom data are or the group to which participants belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): The program with virtual reality will consist of a 30-minutes guided visualization session through virtual reality glasses. Students will visualize a 360º video that simulates the entire experience of an exam, from first person perspective.
  Interventions: Behavioral: Guided visualization of exams through immersive virtual reality
- Experimental group 2 (Active Comparator): The 4-weeks program will consist of a 30-minutes traditional guided visualization session, by listening only the part of the audio used for EG1.
  Interventions: Behavioral: Guided visualization of exams through traditional method
- Control group (No Intervention): This group will not receive any intervention, as the most used strategy to cope with exams among students.

INTERVENTIONS:
Behavioral: Guided visualization of exams through immersive virtual reality — During 4 weeks (twice per week), students will visualize a 30-minutes 360º video that simulates the experience of an exam, from first person perspective.
  Arms: Experimental group 1
Behavioral: Guided visualization of exams through traditional method — During 4 weeks (twice per week), students will listen a 30-minutes audio that explains the experience of an exam from first person.
  Arms: Experimental group 2

SUMMARY:
The new technologies may facilitate the teaching-learning process through the ubiquitous and active approach. However, stress from academic exams remains being high among undergraduate students. Although new technologies could be useful to simulate and control academic stressful situations through immersive virtual reality, no studies to date have evaluated its effectiveness. This study is designed to evaluate the effects of a virtual reality program to visualize stressful academic situations like exams on the level of psychological and physiological stress and academic performance of Physiotherapy and Nursing undergraduate students. To this end, an experimental study with two experimental groups and one control group is designed: experimental group 1 (EG1) will complete a 4-weeks program of guided visualization of exams through immersive virtual reality; experimental group 2 (EG2) will complete a 4-weeks program of traditional guided visualization of exams (through audio); control group (CG) will not receive any visualization program, as the most habitual strategy to cope with exams among students. Before and after the intervention period, all students will fulfill an online questionnaire to inform about their level of academic stress (SISCO inventory) and perceived stress from the last month (Perceived Stress Scale). Also, just before starting the exam they will have been visualizing, level of stress (0 to 10 points), blood pressure (mmHg), maximal heart rate (ppm) and salivary cortisol level will be assessed in all students. Qualifications of the exam will be also collected. Intra-group differences and between-group differences at post-intervention time will be obtained.

DETAILED DESCRIPTION:
As eligibility criteria, participants should be enrolled in at least 80% of subjects of an usual academic course during the year in which the study is carrying out; and not to have previous experience in similar guided visualization to cope with stressful situations.

Intervention of EG1: The 4-weeks program with virtual reality will consist of a 30-minutes guided visualization session through virtual reality glasses (two sessions per week). Students will visualize a 360º video that simulates the entire experience of an exam, from first person perspective.

Intervention of EG2: The 4-weeks program of traditional visualization will consist of a 30-minutes traditional guided visualization session, by listening only the part of the audio used for EG1.

CG will not receive any intervention, as the most used strategy to cope with exams among students. After finishing the study, this group will receive the same program that EG1 or EG2 received, if they are interested.

The main outcomes will be the intra-group and between-group changes in the level of academic stress and the perceived stress from the last month. Also, between-group differences in the level of stress (0 to 10 points), arterial tension (mmHg), maximal heart rate (ppm) and salivary cortisol level just before exams.

As secondary outcomes, between-group differences in qualifications of exams that they will have been visualizing will be also considered (it will be taken into account their average qualifications in the degree).

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in at least 80% of subjects of an usual academic course during the year in which the study is carrying out.
* Not to have previous experience in guided visualization to cope with stressful situations.

Exclusion Criteria:

* Not to understand the Spanish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Academic stress | 4 weeks
  Between-group and intra-group differences in academic stress, which will be registered with the SISCO Inventory version-21. This is the 21-items "Inventario SIStémico COgnoscitivista" for the study of the academic stress, composed by 21 items: the first item is dichotomous (yes-no) and the remaining 20 items are 5-point Likert scale, scored from 1 (never) to 5 (always). The maximal punctuation is 100 (maximal stress).
Perceived stress in the last month | 4 weeks
  Between-group and intra-group differences in perceived stress of the last month, which will be registered with the Perceived Stress Scale. This survey has 10 questions (using Likert scales from 0-5, being 0 never and 5 very often). To interpret this questionnaire, individual scores can range from 0 to 40 with higher scores indicating higher perceived stress.

SECONDARY OUTCOMES:
Level of current perceived stress | Immediately before the exam
  Between-group differences in the level of perceived stress just at the moment prior to start the exam (10 minutes earlier). To evaluate it, students will inform about what level of stress they are feeling at that moment (being 0, no stress, and 10 maximal stress).
Blood pressure | Immediately before the exam
  Between-group differences in the blood pressure just before starting the exam. It will be recorded by a healthcare professional by using a stethoscope and registering the systolic and diastolic blood pressure.
Maximal heart rate | Immediately before the exam
  Between-group differences in the maximal heart rate just before starting the exam
Salivary cortisol level | Immediately before the exam
  Between-group differences in the salivary cortisol level just before starting the exam
Exam qualification (0 to 10 punctuation) pondered by the average qualification of the degree | One week after the exam (an only measurement)
  Between-group differences in the exam qualification (it refers to exam that students will have been visualizing) just before starting the exam. The qualification of the exam will range from 0 (the worst punctuation) to 10 (perfect punctuation). In this outcome, the average qualification of the degree for each student will be considered (from the worst, 0 points, to the best, 10 points). For example, if the student has 8 points as average qualification of the degree and obtains an exam qualification of 9 points, it will be pondered as follows: 9/8 = 1.125.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero-Franco, PhD, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seabrook E, Kelly R, Foley F, Theiler S, Thomas N, Wadley G, Nedeljkovic M. Understanding How Virtual Reality Can Support Mindfulness Practice: Mixed Methods Study. J Med Internet Res. 2020 Mar 18;22(3):e16106. doi: 10.2196/16106. PMID 32186519
- [Result] Riva G, Banos RM, Botella C, Mantovani F, Gaggioli A. Transforming Experience: The Potential of Augmented Reality and Virtual Reality for Enhancing Personal and Clinical Change. Front Psychiatry. 2016 Sep 30;7:164. doi: 10.3389/fpsyt.2016.00164. eCollection 2016. PMID 27746747
- [Result] Lacey C, Frampton C, Beaglehole B. oVRcome - Self-guided virtual reality for specific phobias: A randomised controlled trial. Aust N Z J Psychiatry. 2023 May;57(5):736-744. doi: 10.1177/00048674221110779. Epub 2022 Jul 11. PMID 35818296